CLINICAL TRIAL: NCT05286398
Title: Effect of Cleft Palate Repair Using Alveolar Extension Technique on Primary Dentition and Maxillary Arch Width
Brief Title: Effect of Cleft Palate Repair Using Alveolar Extension Technique on Eruption and Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A09060819
Record Dates: First submitted 2022-03-07; First posted 2022-03-18 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2019-09

CONDITIONS: Cleft Palate
Keywords: Alveolar extension palatoplasty; Bardach; Cleft palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator)
  Interventions: Diagnostic Test: Addition silicone impression
- Bradach group (Experimental)
  Interventions: Procedure: Palatoplasty; Diagnostic Test: Addition silicone impression
- AEP group (Experimental)
  Interventions: Procedure: Palatoplasty; Diagnostic Test: Addition silicone impression

INTERVENTIONS:
Procedure: Palatoplasty — Surgical closure of palatal defect
  Arms: AEP group; Bradach group
Diagnostic Test: Addition silicone impression — diagnostic impression for maxillary arch

SUMMARY:
This study aimed to evaluate clinically the "Alveolar extension" technique for palatoplasty in cases of primary closure of cleft palate regarding its effect on:

1. Eruption of Primary dentition.
2. Maxillary primary teeth undergoing eruption.
3. The maxillary arch growth.

DETAILED DESCRIPTION:
Cleft lip and palate represent the most common of the craniofacial anomalies. They are severe congenital malformations with a worldwide frequency ranging between 0.28 and 3.74 per 1000 live births. Cleft lip and palate occur in around 3 out of every 1000 infants in Egypt. Infants born with cleft palates always have eating difficulties due to a lack of oro-nasal seal and also have speaking difficulties due to velopharyngeal insufficiency. To ensure optimal care, the cleft team may include oral surgeons, plastic surgeons, pediatric dentists, orthodontists, and medical specialists in genetics, otolaryngology, pediatrics, and psychiatry. These caregivers evaluate the medical condition and development of the patient, as well as dental and oral health, facial esthetics, psychological condition, and developing of hearing and speech. Pediatric dentists are critical members of this team because they are responsible for the patient's overall dental health. A variety of dental anomalies and malocclusions are associated with cleft palate; these may occur as a result of primary defects being repaired surgically. The management of the cleft patient starts with an early focus on newborn's needs. Surgical repair of cleft palates (Palatoplasty) is typically performed by one year of age, primarily to facilitate the development of normal speech, as this coincides with the age at which the majority of children begin to speak. Hearing and swallowing are improved by proper alignment of the soft palatal musculature. The ideal palatoplasty technique is one that results in perfect speech without impairing maxillofacial growth or hearing. There are numerous surgical techniques for cleft palate repair, each with numerous variations. Nevertheless, a few of these techniques are widely used. Veau Wardill Kilner Palatoplasty, von Langenbeck, Bardach Two flap Palatoplasty were the most common techniques of palatoplasty. These techniques leave a large raw area along the alveolar margin, exposing bare bone. With secondary intention, the raw area heals. This results in palate shortening and velopharyngeal insufficiency. Additionally, the scar tissue adjacent to the alveolar margin results in deformity of the alveolar ridge and dental malalignment. It was found that lateral incision reduced the maxillary growth more than mucoperiosteal palatal detachment only. Additionally, some studies discovered that when matched normals are compared to individuals with unoperated clefts either lip or palate, the cranial base and skeletal face are not significantly malrelated. These findings suggest that cleft patient possess normal potential and mechanism of growth. The alveolar mucoperiosteum is deprived of blood supply from the facial artery in traditional lip repair procedures. Later, during palate repair, the palatal incisions isolate the palatal tissues from the greater palatine artery, altering the alveolar mucoperiosteum from a highly blood supplied zone between the two arteries into a tissue that is predominantly supported by osseous backflow. Thus, the disruption of palatal growth is considered in this perspective. The Alveolar Extension Palatoplasty (AEP) technique provide tension free flap, less palatal bone exposure after the surgery ,as the raw area is on the alveolar crest or tooth margin. It preserves blood supply of the palatal gingiva and periosteum. The studies on the influence of that advantage as well as the alveolar crest incision on unerupted primary teeth are scanty. So, it will be fruitful to study the effect of AEP on teeth undergoing eruption with alveolar bone and maxilla growth.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes.
2. The age range from 9-12 month.
3. Has a complete cleft palate.
4. Medically fit for general anesthesia.
5. Patients who haven't received any previous palatal repair.

Exclusion Criteria:

1. Syndromic patients.
2. Medically compromised patients contradicting operation.

Ages: 9 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
eruption of primary molars | 6 month
  eruption of primay canine and primary first molar

SECONDARY OUTCOMES:
Growth | 6 monrth
  maxillary arch width

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt